CLINICAL TRIAL: NCT00450775
Title: Evaluation of the Efficacy, Tolerability, and Patient Acceptance of Dermatix Q for the Prevention and Management of Scars
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Innovative Medical (Industry)
Responsible Party: David Rodriguez, MD, Dadeland Dermatology
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 5299
Record Dates: First submitted 2007-03-20; First posted 2007-03-22 (Estimated); Last update posted 2008-09-25 (Estimated); Status verified 2008-09

CONDITIONS: Scars
MeSH Terms: conditions — Cicatrix

ARMS (1):
- 1 (Other)
  Interventions: Drug: Dermatix Q

INTERVENTIONS:
Drug: Dermatix Q — Dermatix Q applied twice daily

SUMMARY:
The purpose of this study is to evaluate the efficacy and patient acceptance of Dermatix Q for the prevention and treatment of scarring.

ELIGIBILITY:
Inclusion Criteria:

* Female or male patients at least 18 years of age
* Patients who are at serious risk of hypertrophic scarring (due to family history, race, recent surgery, etc)
* Able and willing to provide informed consent and likely to complete all study visits
* All Fitzpatrick skin types will be evaluated

Exclusion Criteria:

* Known contraindications to Dermatix or any of its components
* Age of scar is > 4 months
* Keloid scars (scars with increased fibroblastic activity that has exceeded the boundaries of the original scar)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2007-03; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
efficacy | 1 yr

SECONDARY OUTCOMES:
patient acceptance | 1 yr

CONTACTS AND LOCATIONS:
Overall Officials: David Rodriguez, MD, Principal Investigator — Dadeland Dermatology
Locations (1):
- Dadeland Dermatology, Coral Gables, Florida, United States